CLINICAL TRIAL: NCT01305044
Title: Biobehavioral Effects of Tai Chi Chih Among Elderly Female Cancer Survivors
Brief Title: The HEALS Project - Health Education and Active Living for Surviving Seniors
Acronym: HEALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Huntsman Cancer Institute (Other)
Responsible Party: Principal Investigator, Anita Kinney, Professor, Dept of Internal Medicine, University of Utah & Huntsman Cancer Insitute, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 34851; R21 CA135250-2 (Other Grant/Funding Number: NCI); R21CA135250 (NIH)
Record Dates: First submitted 2011-02-18; First posted 2011-02-28 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Cancer Survivorship; Safety and Efficacy; Quality of Life
Keywords: tai chi; elderly cancer survivor; mind body intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tai Chi Chih (Experimental): The Tai Chi Chih classes were 60 minutes sessions, held three times a week, over twelve weeks. The classes were led by an instructor who was certified and licensed in the Tai Chi Chih form.
  Interventions: Behavioral: Tai Chi Chih
- Health Education Classes (Active Comparator): Health Education classes were 60 minute sessions that occurred three times a week, over twelve weeks. These classes were taught by specialists in the class topic and focused on topics related to aging (e.g., sleep quality, nutrition, pain, etc.).
  Interventions: Behavioral: Health Education Classes

INTERVENTIONS:
Behavioral: Tai Chi Chih — Tai Chi Chih (TCC), a westernized and manualized form of the ancient TC Chuan, consists of a series of 20 simple, repetitive, non-strenuous movements that involve no physical contact and emphasize a soft, flowing continuity of motion. This form of meditation through movement consists of a standardized protocol that emphasizes slow, fluid, continuous forms that integrate mental concentration, awareness, balance, shifting of body weight, gentle movement, imagery, muscle relaxation and breathing control. TCC was developed for use with elderly persons.
  Arms: Tai Chi Chih
Behavioral: Health Education Classes — The Health Education classes serve as an attention control group, are led by gerontology specialists, physicians, and other health professionals, and focus on topics that are relevant to elderly cancer survivors.
  Arms: Health Education Classes

SUMMARY:
Persons over age 65 years constitute a large and growing population of cancer survivors. Available data indicate that both short- and long-term female breast cancer survivors report more limitations related to strength and mobility than women with cancers of other sites and women without a personal history of cancer. Further, better mental health among breast cancer survivors has been shown to protect against physical decline and overall quality of life. The combination of mental and physical interventions may result in substantial improvements in quality of life. Tai Chi Chih (TCC), a form of mind-body exercise, is one such intervention. TCC may be particularly suited toward elderly breast cancer survivors with impaired physical and/or mental functioning, yet despite its increasing popularity and benefits in healthy and diseased populations, its benefits have never been scientifically evaluated in this population. The overarching goal of this study is to conduct preparatory work regarding the effects of TCC on quality of life and physical function that will underpin future definitive trials of TCC in elderly cancer survivors. As part of this 12-week trial, participants will be randomized to a TCC or a health education control group (HEC). Establishment of meaningful interventions that facilitate a more positive cancer survival experience in old age is an important issue; there are substantial public health and clinical benefits should a TC intervention be successful in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 55 years and it has been three months or more (with the exception of hormone therapy) since completing treatment for breast or other solid tumor cancers (excluding lung, liver, pancreas and brain) and currently in remission.
2. Living within 30 miles of Huntsman Cancer Institute and has access to transportation and is willing to travel to the study site per study protocol; Travels independently on public transportation or drives own car.
3. Able to speak and read English fluently, and understand informed consent.
4. Willing to: sign a medical record release form; to be randomized and willing to participate in classes and all baseline and follow-up appointments.
5. Has some physical limitation as defined by a score of <72 in the Role Physical or <80 in the Physical Functioning sub-scales in the SF-12 screening questionnaire.
6. Does not currently practice in a regular on-going meditative or relaxation technique.
7. Does not currently engage in a regular, strenuous-intensity form of exercise for 30 min or more per day, 3 or more days per week.

Exclusion Criteria:

1. Engaged in focused intense physical activity for 30 minutes or more a day for 3 or more days a week for the previous 6 months as per responses on the screening telephone call.
2. Regular on-going practice with TC or other similar types of Complementary and Alternative Medicine in the past 6 months such as Qigong, meditation, relaxation, and yoga since these share some of the principles of TC.
3. Inability to pass the Folstein Mini Mental Status Exam (score <23).
4. Unable to drive or secure transportation to complete all aspects of the study.
5. Health conditions (e.g. severe hearing loss, respiratory, cardiovascular, or neurological problems) that might interfere with the required intervention.

Ages: 55 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-12; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kinney, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Result] Campo RA, O'Connor K, Light KC, Nakamura Y, Lipschitz DL, LaStayo PC, Pappas L, Boucher K, Irwin MR, Agarwal N, Kinney AY. Feasibility and acceptability of a Tai Chi Chih randomized controlled trial in senior female cancer survivors. Integr Cancer Ther. 2013 Nov;12(6):464-74. doi: 10.1177/1534735413485418. Epub 2013 Apr 25. PMID 23620504

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 371 female cancer survivors with some functional limitations were recruited through Huntsman Cancer Institute registries and clinics, and community advertisements (media, newspapers). The first cohort of participants was held in the Spring 2010 with the second and third cohorts of participants held in the Fall 2010 and Spring 2011, respectively.
Pre-assignment Details: Forty percent (n=150) expressed an interest in participating and 42% who met eligibility (n=63) were randomized to receive 12-week (3 days/week) of TCC or Health Education Control (HEC) classes.
Groups:
- Tai Chi Chih: Tai Chi Chih : Tai Chi Chih (TCC), a westernized and manualized form of the ancient TC Chuan, consists of a series of 20 simple, repetitive, non-strenuous movements that involve no physical contact and emphasize a soft, flowing continuity of motion. This form of meditation through movement consists of a standardized protocol that emphasizes slow, fluid, continuous forms that integrate mental concentration, awareness, balance, shifting of body weight, gentle movement, imagery, muscle relaxation and breathing control. TCC was developed for use with elderly persons.
- Health Education: Health Education Classes : The Health Education classes serve as an attention control group, were led by gerontology specialists, physicians, and other health professionals, and focus on topics that are relevant to elderly cancer survivors.
Period: Overall Study
Arm/Group | Tai Chi Chih | Health Education
Started | 32 | 31
Completed | 29 | 25
Not Completed | 3 | 6
Not completed — Withdrawal by Subject | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tai Chi Chih | Health Education | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 20 | 19 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 31 | 63

OUTCOME MEASURES:

1. Primary Outcome: Retention Rates and Class Attendance
Description: The 12-week intervention assessed retention in the study (percentage of how many participants remained enrolled the entire intervention), class attendance (percentage out of possible classes)
Time Frame: 13 weeks
Population: Power calculations indicated that a sample size of 42 would be sufficient to detect 15 point change in SF-36, with 88% power at 5% significance level. Analysis were per protocol because the sample size was too small for imputation techniques and there was no follow-up data on withdrawn participants for intent-to-treat analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Tai Chi Chih | Health Education
Number analyzed (Participants) | 29 | 25
percentage of participants
  Retention Rate | 91 | 81
  Class Attendance Rate | 79 | 83

2. Secondary Outcome: Health-Related Quality of Life (Short Form (SF)-36v1)
Description: SF-36v1 Health Survey assesses quality of life and produces mental and physical component summary scores, with a score range of 0 to 100. Higher scores indicate better quality of life.
Time Frame: 13 weeks
Population: Please refer to power calculation detailed in Primary Outcome Measure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Tai Chi Chih | Health Education
Number analyzed (Participants) | 29 | 25
units on a scale
  Mental Component Summary Score | 51.7 (1.6) | 51.0 (1.6)
  Physical Component Summary Score | 41.3 (1.4) | 43.2 (1.5)

3. Secondary Outcome: Perceived Stress Scale
Description: The 10-item perceived stress scale produces a summation score. Scores can range from 0 to 40, with higher scores indicating more stress.
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tai Chi Chih | Health Education
Number analyzed (Participants) | 29 | 25
units on a scale | 12.0 [5.0 to 17.0] | 13.0 [7.0 to 17.0]

4. Secondary Outcome: Impact of Events Scale
Description: The Impact of Event Scale assesses cancer-specific distress. Each item is scored 0 (not at all), 1 (rarely), 3 (sometimes)or 5 (often), with the higher scores reflecting more stressful impact. It has a total score and two subscales (avoidance & intrusion). The two subscales are scored by summing their corresponding items and the total score is the sum of two subscales. The scores for the intrusive subscale range from 0 to 35, and scores for the avoidance subscale range from 0 to 40. The Total Score ranges from 0-75, with higher scores reflecting more stressful impact.
Time Frame: 13-weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tai Chi Chih | Health Education
Number analyzed (Participants) | 29 | 25
units on a scale
  Total Score | 22.0 [18.0 to 26.0] | 19.0 [15.0 to 28.0]
  Avoidance Subscale | 13.0 [11.0 to 17.0] | 11.0 [8.0 to 14.0]
  Intrusion Subscale | 10.0 [7.0 to 11.0] | 9.0 [7.0 to 10.0]

5. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: The Pittsburgh Sleep Quality produces a global score. The range is 0 to 21, higher scores indicate worse sleep quality.
Time Frame: 13-weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tai Chi Chih | Health Education
Number analyzed (Participants) | 29 | 25
units on a scale | 8.0 [6.0 to 11.0] | 10.0 [7.0 to 11.0]

6. Secondary Outcome: Five-Facet Mindfulness Questionnaire
Description: The Five-Facet Mindfulness questionnaire produces a total score and five facet subscales (observing, describing, acting with awareness, nonjudging, & nonreactivity). These are summation scores, and the scores range from 8 to 40 (except for the nonreactivity facet which ranges from 7 to 35). Higher scores indicate more mindfulness. The Total Score ranges from 39-195, with higher scores indicating more mindfulness.
Time Frame: 13-weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tai Chi Chih | Health Education
Number analyzed (Participants) | 29 | 25
units on a scale
  Total Mindfulness Score | 125.0 [108.2 to 137.8] | 136.5 [114.5 to 152.2]
  Observing Subscale | 28.0 [16.0 to 32.0] | 29.0 [25.0 to 35.0]
  Describing Subscale | 26.0 [23.0 to 30.0] | 30.0 [24.0 to 34.0]
  Awareness Subscale | 20.0 [16.0 to 22.0] | 22.0 [17.0 to 26.0]
  Nonjudging Subscale | 24.0 [17.0 to 30.0] | 28.5 [24.7 to 31.2]
  Nonreacting Subscale | 25.5 [21.7 to 29.0] | 25.0 [21.0 to 29.0]

7. Secondary Outcome: Blood Pressure
Description: Systolic and Diastolic blood pressure were assessed at the study's physical assessment sessions.
Time Frame: 13-weeks
Population: Please refer to power calculation detailed in Primary Outcome Measure.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Tai Chi Chih | Health Education
Number analyzed (Participants) | 29 | 25
mm Hg
  Systolic Blood Pressure | 119.0 (2.8) | 132.5 (3.1)
  Diastolic Blood Pressure | 79.6 (2.2) | 79.7 (2.4)

8. Secondary Outcome: Cortisol Area-Under-Curve (AUC)
Description: Five saliva samples (awakening, 30 minutes after awakening, noon, 5pm, & 10pm) were collected on a weekend day at one week after class completion. Cortisol was measured in nmol/L. Cortisol AUC was calculated using the five timepoints with the trapezoid rule. The groups were compared at post-intervention on their log transformed cortisol AUC controlling for baseline cortisol and reported as adjusted means. Four participants with high cortisol profiles across the five collection times (with suspected contamination from gum bleeding) and participants whose collection time was beyond a one hour window were excluded.
Time Frame: 13-weeks
Measure: Mean (Standard Error); unit: nmol*hr/L
Arm/Group | Tai Chi Chih | Health Education
Number analyzed (Participants) | 20 | 19
nmol*hr/L | 24.6 (1.5) | 29.9 (1.5)

9. Secondary Outcome: Inflammatory Cytokines
Description: Fasting blood samples were collected in the morning for inflammatory cytokines. Prior to blood draws, we ensured that participants did not experience illness or fever at the time of the blood draw. The assayed cytokines included pro-inflammatory cytokines interleukin(IL)-12, IL-6, tumor necrosis factor (TNF)-α, and anti-inflammatory cytokines IL-10 and IL-4.
Time Frame: 13-weeks
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Tai Chi Chih | Health Education
Number analyzed (Participants) | 28 | 24
pg/ml
  IL-12 | 4.7 [3.3 to 12.5] | 3.7 [1.3 to 7.4]
  IL-6 | 9.1 [4.3 to 29.0] | 5.3 [3.4 to 8.2]
  TNF-α | 37.8 [0 to 77.9] | 45.1 [0 to 109.1]
  IL-4 | 1.5 [0.6 to 3.6] | 1.1 [0.5 to 2.2]
  IL-10 | 5.8 [4.3 to 16.3] | 5.0 [2.9 to 7.7]

10. Primary Outcome: Satisfaction With the Randomized Controlled Trial
Description: The 12-week intervention assessed satisfaction with intervention(0=strongly agree to 4=strongly disagree).
Time Frame: 13 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tai Chi Chih | Health Education
Number analyzed (Participants) | 29 | 25
units on a scale | 1.00 [.78 to 1.2] | 1.11 [1.00 to 1.6]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Tai Chi Chih | Health Education
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No